CLINICAL TRIAL: NCT02071277
Title: Impact of the Type of Pressure Controlled Mode on Lung Protection in Mechanically Ventilated Patients With Spontaneous Breathing
Brief Title: APRV/BIPAP With Spontaneous Breathing on Lung Protection
Acronym: APRV/BIPAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Unity Health Toronto (Other)
Collaborators: University of Toronto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: REB 13-362
Record Dates: First submitted 2014-02-07; First posted 2014-02-25 (Estimated); Last update posted 2017-04-19 (Actual); Status verified 2017-04

CONDITIONS: Respiratory Insufficiency; Ventilator-Induced Lung Injury
Keywords: Mechanical ventilation; Airway pressure release ventilation; Biphasic intermittent positive airway pressure; Pressure-controlled ventilation; Lung protective ventilation; Spontaneous breathing
MeSH Terms: conditions — Respiratory Insufficiency; Ventilator-Induced Lung Injury

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Pressure targeted modes (Experimental)
  Interventions: Other: Pressure targeted modes

INTERVENTIONS:
Other: Pressure targeted modes — Intervention involving three different pressure-targeted modes (APRV, BIPAP, and BIPAPassist) each in a random order generated by a computer on one ventilator. Each mode will be studied for 20 minutes.

SUMMARY:
Mechanical ventilation (MV) is a cornerstone of management of acute respiratory failure, but MV per se can provoke ventilator-induced lung injury (VILI), especially in acute respiratory distress syndrome (ARDS). Lung protective ventilation strategy has been proved to prevent VILI by using low tidal volume of 6-8 ml/kg of ideal body weight and limiting plateau pressure to less than 30 cmH2O. However, heavy sedation or even paralysis are frequently used to ensure the protective ventilation strategy, both of which are associated with respiratory muscles weakness. Maintaining of spontaneous breathing may decrease the need of sedative drug and improve gas exchange by promoting lung recruitment.

Pressure-targeted mode is the most frequent way of delivering after 48 hours of initiating MV. Three types of pressure-controlled mode are available in intubated patients: Biphasic Intermittent Positive Airway Pressure (BIPAP), Airway Pressure Release Ventilation (APRV), and Pressure-Assist Controlled Ventilation (also called BIPAPassist). They are based on pressure regulation but have the difference in terms of synchronization between the patient and the ventilator. The different working principle of these modes may result in different breathing pattern and consequently different in tidal volume and transpulmonary pressure, which may be potentially harmful. The investigators bench study with a lung model demonstrated higher tidal volume and transpulmonary pressure with the BIPAPassist over APRV despite similar pressure settings and patient's simulated effort. However, the impact of each mode on the delivered tidal volume and the transpulmonary pressure in spontaneously breathing mechanically ventilated patients is currently unknown. Their hypothesis is that when the investigators compare the three pressure-controlled modes, the asynchronous mode (APRV) will result in more protective ventilation strategy over the two other modes (BIPAP and BIPAPassist).

ELIGIBILITY:
Inclusion Criteria: Patients who admitted in the intensive care unit (ICU) and mechanically ventilated (through an endotracheal or a tracheostomy tube) and meet the following criteria are eligible for study participation:

* Male or female patient,
* Age over 18 years,
* Patient already ventilated with assist controlled mode (volume or pressure) and patient triggering the ventilator,
* Arterial line indwelling or planning to insert this line,
* Written informed consent signed and dated by the patient/next of kin after full explanation of the study by the study team and prior to study participation,
* Patient consent will be requested as soon as the patient will be able to provide informed written consent

Exclusion Criteria: Patients who fulfill any of the following exclusion criteria are not eligible for study participation:

* Hemodynamic instability
* > 20% variation of mean arterial pressure and/or heart rate (HR) in the last 2 hours,
* Need for high dose of vasopressor (higher than 0.2 mcg/kg/min of levophed),
* High PEEP (> 12 cmH2O) and/or high fraction of inspired oxygen inspired oxygen fraction (> 0.6)
* Severe acidosis (pH ≤ 7.20), or severe alkalosis (pH > 7.55)
* Presence of a known esophageal problem, active upper gastrointestinal bleeding or any other contraindication to the insertion of a oro- or naso-gastric tube,
* Pregnant patient,
* Presence of intracranial hypertension,
* Known chronic neuromuscular disease significantly impairing the spontaneous breathing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2014-03; Primary Completion 2017-01 (Actual); Study Completion 2017-03-15 (Actual)

PRIMARY OUTCOMES:
Tidal volume in each mode of ventilation | 20 minutes

SECONDARY OUTCOMES:
Inspiratory transpulmonary pressure in each mode of ventilation | 20 minutes
Patient work of breathing | 20 minutes
  Patient work of breathing will be measured by using pressure-time product and pressure generated 100 ms after the onset of an occluded inspiratory effort (P0.1)
The frequency of each breath-type according to the mode | 20 minutes
  Type A: spontaneous breaths occurring during Tlow, Type B: spontaneous breaths occurring during Thigh, Type C: quasi-assisted breaths synchronized with the ventilator cycling to Thigh, Type D: completely passive breaths, Type E: spontaneous breaths occurring as the ventilator cycles to Tlow

CONTACTS AND LOCATIONS:
Overall Officials: Laurent Brochard, Dr., Principal Investigator — Unity Health Toronto
Locations (2):
- Canada (2):
  - St. Michael's Hospital, Toronto, Ontario
  - Mount Sinai Hospital, Toronto, Ontario

REFERENCES:
- [Background] Richard JC, Lyazidi A, Akoumianaki E, Mortaza S, Cordioli RL, Lefebvre JC, Rey N, Piquilloud L, Sferrazza Papa GF, Mercat A, Brochard L. Potentially harmful effects of inspiratory synchronization during pressure preset ventilation. Intensive Care Med. 2013 Nov;39(11):2003-10. doi: 10.1007/s00134-013-3032-7. Epub 2013 Aug 9. PMID 23928898
- [Derived] Rittayamai N, Beloncle F, Goligher EC, Chen L, Mancebo J, Richard JM, Brochard L. Effect of inspiratory synchronization during pressure-controlled ventilation on lung distension and inspiratory effort. Ann Intensive Care. 2017 Oct 6;7(1):100. doi: 10.1186/s13613-017-0324-z. PMID 28986852